CLINICAL TRIAL: NCT04382911
Title: Evaluation of Endometriosis With 18F-fluoroestradiol PET / MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-0328
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-fluoroestradiol PET / MRI (Experimental): All enrolled subjects will receive the tracer and then have a PET/MRI scan.
  Interventions: Drug: 18F-fluoroestradiol

INTERVENTIONS:
Drug: 18F-fluoroestradiol — Patients will receive the FES tracer during a PET/MRI scan
  Other Names: FES

SUMMARY:
Purpose: The primary objective is to evaluate the sensitivity and specificity of 18F-fluoroestradiol (FES) PET/MRI for evaluating endometriosis.

Participants: A total of 12 participants will be recruited from individuals with clinically suspected endometriosis who are scheduled for planned operative laparoscopy at the University of North Carolina at Chapel Hill (UNC).

Procedures (methods): This is a prospective, one arm, single center study of 12 subjects with clinically suspected endometriosis to demonstrate FES PET/MR's clinical utility for diagnosis of endometriosis. This study will be an evaluation of the radiotracer, FES, which binds to estrogen receptors and has previously been used to study estrogen receptor expression in tumors, to detect endometriosis. Participants will undergo one FES PET/MR scan within 4 weeks prior to their scheduled surgery. Participants will also complete questionnaires regarding their condition, pain, and quality of life.

DETAILED DESCRIPTION:
This is a prospective, one arm, single center study of 12 subjects with clinically suspected endometriosis to demonstrate FES PET-MRI's clinical utility for diagnosis of endometriosis. The primary objective is to evaluate the sensitivity and specificity of 18F-fluoroestradiol (FES) PET/MRI for evaluating endometriosis. Secondary objectives include comparing PET to conventional MRI, using histopathology from laparotomy as the gold standard and evaluating association of uptake values (SUV-max) with Endometriosis Health profile -30 (EHP-30) and pain rating scales, controlling for covariates.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Female of childbearing age
* Clinically suspected (symptomatic) endometriosis.
* Scheduled for planned operative laparoscopy with no hormone treatment for at least two cycles
* Able to provide informed consent or assent

Exclusion Criteria:

* Male
* Institutionalized subject (prisoner or nursing home patient)
* Known history of breast, ovarian or endometrial cancer.
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Oldan, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-fluoroestradiol PET / MRI: All enrolled subjects will receive the tracer and then have a PET/MRI scan. A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan.
  18F-fluoroestradiol (FES): Patients will receive 6 mCi of the FES tracer during a PET/MRI scan
Period: Overall Study
Arm/Group | 18F-fluoroestradiol PET / MRI
Started | 8
Completed | 6
Not Completed | 2
Not completed — unable to be imaged prior to surgery | 2

BASELINE CHARACTERISTICS:
Groups:
- 18F-fluoroestradiol PET / MRI: All enrolled subjects will receive the tracer and then have a PET/MRI scan. A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan
  18F-fluoroestradiol: Patients will receive the FES tracer during a PET/MRI scan
Arm/Group | 18F-fluoroestradiol PET / MRI
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Pain Rating Scales (Visual Analog Scale - VAS) [Mean (Standard Deviation); unit: mm] — Individuals will be given a 100mm scale and asked to draw a single vertical line corresponding to the level of pain where 0mm is no pain and 100mm is pain as bad as it possibly could be. This line will be measured and the result will be recorded in mm. Population: One participant did not complete the VAS questionnaire.
  mm
    number analyzed (Participants) | 7
    (all) | 11.71 (25.06)
Endometriosis Health Profile-30 (EHP-30) [Mean (Standard Deviation); unit: units on a scale] — The Endometriosis Health Profile-30 (EHP-30), a quality of life questionnaire used in women with endometriosis, includes questions related to pain, control and powerlessness, social support, emotional wellbeing, and self-image. Each scale is standardized on a scale of 0 - 100, where 0 indicates the best health status through to 100 worst health status. Scale scores for each scale are calculated from the total of the raw scores of each item in the scale divided by the maximum possible raw score of all the items in the scale, multiplied by 100. Population: One participant did not complete the EHP-30 questionnaire
  units on a scale
    number analyzed (Participants) | 7
    (all) | 40.7 (28.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a person's weight in kilograms (or pounds) divided by the square of height in meters (or feet).
  kg/m^2 | 26.54 (4.81)

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of FES PET/MRI for Evaluating Endometriosis (Percentage of Positive Scans)
Description: The sensitivity of FES PET /MRI is defined as the ability of readers (radiologists) to detect endometriosis among those with histopathologically identified endometriosis in the entire cohort. Sensitivity is calculated by dividing the number of true cases of endometriosis by the overall number of patients with endometriosis identified using the research imaging. The sensitivity data can only be calculated upon completion of study imaging for all participants.
Time Frame: day of scan, up to 2 hours
Population: Two of the 8 enrolled subjects were unable to be imaged and therefore are not included in the analysis.
Measure: Number; unit: percentage of positive scans
Units Other Than Participants: scans
Groups:
- 18F-fluoroestradiol PET / MRI: All enrolled subjects will receive the tracer and then have a PET/MRI scan. A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan.
  18F-fluoroestradiol: Patients will receive the FES tracer during a PET/MRI scan.
Arm/Group | 18F-fluoroestradiol PET / MRI
Number analyzed (Participants) | 6
Number analyzed (scans) | 6
percentage of positive scans | 67
Statistical Analysis 1: Comparison: 18F-fluoroestradiol PET / MRI; Test type: Equivalence — A 2x2 table was constructed among all patients with histopathologically identified endometriosis (true positive) to compare sensitivity for FES PET/MRI versus sensitivity of conventional MRI; p = 0.317, McNemar

2. Primary Outcome: Specificity of FES PET/MRI for Evaluating Endometriosis (Percentage of Negative Scans)
Description: The specificity of FES PET /MRI is defined as the ability of readers (radiologists) to detect that patients do not have endometriosis divided by the number of participants without endometriosis as defined histopathologically in the entire cohort. Specificity is calculated by dividing the number of true negative cases by the overall number of patients without endometriosis identified using the research imaging. The specificity data can only be calculated upon completion of study imaging for all participants.
Time Frame: day of scan, up to 2 hours
Population: The specificity is undefined since the denominator is 0 as all participants had endometriosis.
Arm/Group | 18F-fluoroestradiol PET / MRI
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of the FES PET/MRI Specificity to Conventional MRI
Description: The investigators will use McNemar's test, constructing the 2x2 table among all patients with a surgical diagnosis of negative to compare specificity for FES PET/MRI (Outcome Measure 2) versus conventional MRI. The specificity of FES PET /MRI is defined as the ability of readers (radiologists) to detect that patients do not have endometriosis divided by the number of participants without endometriosis as defined histopathologically in the entire cohort. Specificity is calculated by dividing the number of true negative cases by the overall number of patients without endometriosis identified using the research imaging. The specificity data can only be calculated upon completion of study imaging for all participants.
Time Frame: day of scan, up to 2 hours
Population: The specificity is undefined since the denominator is 0 as all participants had endometriosis.
Arm/Group | 18F-fluoroestradiol PET / MRI
Number analyzed (Participants) | 0

4. Secondary Outcome: Mean Standard Uptake Values (SUV-max) for 18F-fluoroestradiol PET / MRI
Description: The SUV-max is the maximum standardized uptake value for FES within the tissue.
Time Frame: day of scan, up to 2 hours
Population: Two of the eight enrolled subjects were unable to be imaged and therefore are not included in the analysis because SUV-max can only be determined using the research scan.
Measure: Mean (Standard Deviation); unit: SUV-max
Units Other Than Participants: scans
Arm/Group | 18F-fluoroestradiol PET / MRI
Number analyzed (Participants) | 6
Number analyzed (scans) | 6
SUV-max | 3.23 (3.04)
Statistical Analysis 1: Comparison: 18F-fluoroestradiol PET / MRI; Test type: Other — A random effects linear regression model, modeling SUV-max as a function of the pain rating, while controlling for patient-level covariates (BMI, race, age) was performed. The investigators included physician as a random effect to account for physician-level correlation; p = 0.24, Pearson's Correlation Coefficient; Slope = 0.748
Statistical Analysis 2: Comparison: 18F-fluoroestradiol PET / MRI; Test type: Other — The investigators will implement a random effects linear regression model, modeling SUV-max as a function of EHP-30, while controlling for patient-level covariates (BMI, race, age). The investigators will include physician as a random effect to account for physician-level correlation; p = 0.13, Mixed Models Analysis; Slope = 0.406

ADVERSE EVENTS:
Time Frame: Assessed for 24 hours following the imaging procedure.
Arm/Group | 18F-fluoroestradiol PET / MRI
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-fluoroestradiol PET / MRI (N=6)
Fatigue (General disorders) | 1 (1) — Patient reported fatigue lasting 4 hours following the procedure.
Change in smell (General disorders) | 1 (1) — Subject reported change in smell for 4 hours, which was determined to be unrelated.
headache (General disorders) | 1 (1) — Patient reported a headache that resolved, which was determined to be unrelated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT04382911/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04382911/ICF_001.pdf